CLINICAL TRIAL: NCT03917979
Title: Effectiveness of the Bonny Method of Guided Imagery and Music (GIM) in the Treatment of Depression: A Randomized Controlled Trial
Brief Title: The Bonny Method of Guided Imagery and Music (GIM) in the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Appalachian State University (Other)
Responsible Party: Principal Investigator, Tim Honig, PhD Researcher, Doctoral Programme in Music Therapy, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIM Depression
Record Dates: First submitted 2019-04-13; First posted 2019-04-17 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: Music Therapy; Guided Imagery; Randomized Controlled Trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is not possible to fully mask participants to the treatment they receive since they will know whether their sessions start immediately or after 20 weeks and whether their sessions are individual or in a group. Similarly, it is not possible to mask the care provider to the participants' condition. However, participants will be masked to which condition is the experimental condition and which is the control condition, and all will receive a series of GIM sessions either in groups or as individuals. The outcome assessors will be masked to participants' group assignment during data collection since participants will complete data collection procedures by mailed packet of self-report measures. All self-report packets will be identified only by a unique client number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual GIM (Experimental): Participants are provided with a series of individual GIM sessions.
  Interventions: Behavioral: Individual GIM
- Waitlist Control (Other): Participants complete an initial wait list period, then are provided with a series of Group GIM sessions.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Individual GIM — Participants are provided with a series of 10 individual GIM sessions, scheduled once every two weeks. Frequency may change if clinically indicated. Individual GIM sessions begin with a discussion of important issues related to the client's life and symptoms, forming a focus for the session. Then, the therapist provides suggestions to help the client become highly relaxed and focused in preparation for the music-listening portion of the session. The therapist plays specially-selected music from the Western classical tradition to match the client and the focus for the session, and engages in verbal dialogue with the client to help them explore their own internal imagery while listening to the music. After the music ends, the therapist and client engage in discussion about their imagery in metaphoric connection to their therapeutic process. This may include arts-based approaches to process the session. Sessions last approximately 90-120 minutes.
  Arms: Individual GIM
Behavioral: Waitlist Control — Participants complete an initial wait list period of 26 weeks, equivalent to the treatment and 6-week follow-up period for the experimental arm. They are then provided with four Group GIM sessions scheduled once per week. Group GIM sessions start with a group discussion about events or feelings from the week and issues related to depression and wellbeing. Then the therapist provides suggests to help the clients relax and focus in preparation for the music-listening period. Group members will explore a theme or issue related to therapy while focusing on whatever comes to them as the music is played. After the music, there will be a time to work with the imagery experienced during the music. This may be in the form of discussion or other art forms. The session ends with a discussion about gains and insights from the music and imagery. Sessions last 90-120 minutes.
  Arms: Waitlist Control

SUMMARY:
The purpose of this research is to study the effectiveness of the Bonny Method of Guided Imagery and Music (GIM) as a treatment approach for depression. Specifically, this study will examine the treatment outcomes of a series of individual GIM sessions for persons with mild or moderate depression. It is guided by the following three research questions: In individuals with depression, does a series of GIM sessions 1) reduce severity of depression, 2) reduce severity of anxiety, and 3) improve mental well-being in comparison to a control group? The hypothesis is that a series of individual GIM sessions will be associated with improvement in depression, anxiety, and mental well-being that is greater than the waitlist control group.

GIM is a music-centered integrative therapy approach. In it, therapist-selected programs of music from the Western classical tradition are used to evoke and develop a client's spontaneously generated imagery in a highly focused non-ordinary state of consciousness. In dialogue with the therapist, the client explores this imagery in a metaphoric, transformative process.

After providing informed consent and verifying that they meet all eligibility requirements, 30 participants are randomly assigned to either a treatment condition or waitlist control condition. Participants in the treatment group are provided with a series of 10 individual GIM sessions occurring once every two weeks. Individuals in the waitlist condition are provided with a series of four Group GIM sessions after the initial waitlist period. All participants complete data collection packets at pre-test, midpoint, posttest, 6-week follow-up, and 12-week follow-up.

The individual and group GIM sessions are conducted by board-certified music therapists (MT-BC) who have completed training in the Bonny Method of Guided Imagery and Music and have the credential Fellow of the Association for Music and Imagery (FAMI). The researchers will implement a Quality Assurance protocol to monitor fidelity to treatment.

GIM is a therapeutic approach accessible on a limited basis worldwide, and trained practitioners are granted credentials by the Association for Music and Imagery (AMI) and Music and Imagery Association of Australia (MIAA). Databases of practitioners are available through these organizations.

DETAILED DESCRIPTION:
The purpose of this research is to study the effectiveness of the Bonny Method of Guided Imagery and Music (GIM) as a treatment approach for depression. Specifically, this study will examine the treatment outcomes of a series of individual GIM sessions for persons with mild or moderate depression. It is guided by the following three research questions: In individuals with depression, does a series of GIM sessions 1) reduce severity of depression, 2) reduce severity of anxiety, and 3) improve mental well-being in comparison to a control group? The hypothesis is that a series of individual GIM sessions will be associated with improvement in depression, anxiety, and mental well-being that is greater than the waitlist control group.

Background: The Bonny Method of Guided Imagery and Music is a music-centered depth approach to exploring the self. In GIM, therapist-selected programs of music from the Western classical tradition are used to evoke and develop a client's spontaneously generated imagery in a highly focused non-ordinary state of consciousness. In dialogue with the therapist, the client explores this imagery in a transformative process.

Preliminary evidence suggests that the Bonny Method of Guided Imagery and Music may be an appropriate therapeutic approach for persons with depression. Used in psychotherapy, it has been documented as treatment for depression in qualitative research, case studies and clinical practice. There is quantitative evidence that GIM may be effective at reducing depression and related symptoms in a variety of clinical and nonclinical populations. A systematic review examined the evidence of psychological and physiological change associated with a series of individual GIM sessions and found a cluster of positive treatment effects related to mood including improvements in depression and depressed mood, mood disturbance, and anxiety. There is also evidence that these treatment effects may persist over time.

Design: This quantitative research will use a split-plot factorial, or mixed, design with two conditions: (a) an experimental group who receive a series of individual GIM sessions and (b) a waitlist control group who receive a series of group GIM sessions after completing a waitlist period. The research is utilizing a waitlist control condition to meet the ethical demand of providing a degree of parity between experimental and control condition, improve feasibility of the research, and to mitigate bias produced by the inability to fully mask participants to their group assignment. The research will be conducted in a naturalistic setting in a private office in a psychology and counseling practice that has been retained for the length of the research study. This research is studying intervention effectiveness rather than efficacy, and therefore the design allows for a degree of flexibility with the provision of the intervention as is normal in a real-world clinical setting.

Recruitment: Adults seeking treatment for depression will be recruited from outpatient mental health care providers and from the community. At the time of enrollment in the study, participants will be asked to provide the name and contact information of their most recent mental health care provider. In the event that a participant requires more intensive treatment while participating in the research study, the participant will be referred to that mental health care provider for a formal assessment. If a participant does not provide information for a mental health care provider, they will be referred to a mental health assessment and referral center in the community.

Randomization: After providing informed consent and verifying that they meet all eligibility requirements, participants are randomly assigned to either a treatment condition or waitlist control condition. The study will use block randomization to ensure even group allocation at both clinical sites, and will be conducted by a member of the research team who is not involved in recruitment, screening, or providing the intervention.

Clinical Sites: Clinical sessions for the study will take place at two research sites in the United States: one metropolitan area in the Midwest and one in the mid-Atlantic. The individual and group GIM sessions will be conducted by board-certified music therapists (MT-BC) who have completed training in the Bonny Method of Guided Imagery and Music as endorsed by the Association for Music and Imagery, and have the credential Fellow of the Association for Music and Imagery (FAMI).

Quality Assurance: To ensure consistent and high-quality treatment and maximize internal and external validity, the research team will monitor fidelity to the GIM approach in each session with a GIM Treatment Fidelity Assessment, created for the purposes of this research. This assessment will be completed by the therapist immediately following each GIM session. Any signs of variation, drift, or bias will be discussed with the research team. The therapists will also receive clinical supervision from an experienced GIM supervisor throughout the course of the study. All sessions will be audio-recorded for reference related to quality assurance.

Data Collection: All participants complete data collection packets at pre-test, midpoint (week 10), posttest (week 20), 6-week follow-up, and 12-week follow-up. Based on power calculations using effect size estimates (d = 0.5) from previous research, the study is seeking a total of 30 participants, adjusted to include an additional 20% to account for attrition. At each time point, participants will complete self-report measures related to depression, anxiety, and mental well-being, and give information about changes in other therapies or medical treatment. Because this is the first randomized controlled trial (RCT) examining GIM in the treatment of depression, the study is not controlling access to other therapies or medical care while participants are involved in the study. However, information on other therapies or medical care will be collected at all data points to allow the researchers to assess the degree to which these factors may have biased the results in the final analysis.

Data Analysis: In the case of attrition or missing data, statistical analysis will utilize the intent-to-treat principle. Data analysis will be conducted using Statistical Package for the Social Sciences (SPSS) and analyzed according to the split-plot factorial design. The factors are 1) treatment group and 2) time. Factor 1 has two levels: GIM and waitlist control. Factor 2 has four levels: pretest, midpoint, posttest, and 6-week follow-up. Note that the 12-week follow-up will not be included in the main data analysis because the waitlist control group will have received Group GIM during that period. A secondary repeated measures analysis of the experimental group will be undertaken to examine the 12-week follow-up data.

The data will first be examined to test the assumptions for parametric statistics with split-plot factorial ANOVA. If the data do not meet these assumptions, the data will be analyzed using aligned rank-transformation. Once aligned and rank-transformed, the data will be analyzed using split-plot factorial ANOVA.

If the data do meet the assumptions for parametric statistics, the data will be analyzed using split-plot factorial ANOVA. In the case of a nonsignificant or ordinal interaction, main effects will be examined. In the case of a significant disordinal interaction, a simple effects analysis will be completed for time within-subjects. In the case of significant change in any of the dependent variables over time, post hoc analyses will be conducted to determine between which time points the significant change occurred. Effect sizes (Cohen's d) and confidence intervals will be calculated and reported for all outcomes, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or over
* Meet severity threshold for mild to moderate depression as measured by the Inventory of Depressive Symptomatology (IDS-SR; score of 14-38) at the time of enrollment
* English-speaking
* Able to read and write at a fifth grade level or higher

Exclusion Criteria:

* History of psychosis
* Diagnosis related to depression other than unipolar depression, including but not limited to bipolar disorder and schizoaffective disorder
* Meeting threshold for severe depression as measured by the Inventory of Depressive Symptomatology (IDS-SR; score greater than 38) at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Depression score as measured by the IDS-SR | Pretest at the time of enrollment, midpoint (week 10), posttest (week 20), 6-week follow-up (week 26), 12-week follow-up (week 32)
  Mean change in total score (range of 0-84) for the Inventory of Depressive Symptomatology - Self-report (IDS-SR). Change is assessed among all time points. A higher score represents greater severity of depressive symptoms, and a lower score represents a better outcome.
Mean change from baseline in Depression score as measured by the Depression, Anxiety, and Stress Scales (DASS) | Pretest at the time of enrollment, midpoint (week 10), posttest (week 20), 6-week follow-up (week 26), 12-week follow-up (week 32)
  Mean change in total score for the depression scale of the DASS. Scores for the depression scale range from 0-42. A higher score represents greater severity of depression and a worse outcome, and a lower score represents reduced depressive symptoms and a better outcome. Change is assessed among all timepoints.
Mean change from baseline in Anxiety score as measured by the Depression, Anxiety, and Stress Scales (DASS) | Pretest at the time of enrollment, midpoint (week 10), posttest (week 20), 6-week follow-up (week 26), 12-week follow-up (week 32)
  Mean change in total score for the Anxiety scale of the DASS. Scores for the Anxiety scale range from 0-42. A higher score represents greater severity of anxiety and a worse outcome, and a lower score represents a better outcome. Change is assessed among all timepoints.
Mean change from baseline in mental well-being score as measured by the WEMWBS | Pretest at the time of enrollment, midpoint (week 10), posttest (week 20), 6-week follow-up (week 26), 12-week follow-up (week 32)
  Score for the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS). Change is assessed among all timepoints.

SECONDARY OUTCOMES:
Mean change from baseline in Stress score, as measured by the Depression, Anxiety, and Stress Scales (DASS) | Pretest at the time of enrollment, midpoint (week 10), posttest (week 20), 6-week follow-up (week 26), 12-week follow-up (week 32)
  Mean change in total score for the Stress scale of the DASS. Scores for the Stress scale range from 0-42. A higher score represents greater severity of stress and a worse outcome, and a lower score represents a better outcome. Change is assessed among all timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Honig, MMT, Principal Investigator — Aalborg University
Locations (2):
- United States (2):
  - Guided Imagery and Music Research, Westfield, Massachusetts
  - Guided Imagery and Music Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borrelli B. The Assessment, Monitoring, and Enhancement of Treatment Fidelity In Public Health Clinical Trials. J Public Health Dent. 2011 Winter;71(s1):S52-S63. doi: 10.1111/j.1752-7325.2011.00233.x. PMID 21499543
- [Background] Chou MH, Lin MF. Exploring the listening experiences during guided imagery and music therapy of outpatients with depression. J Nurs Res. 2006 Jun;14(2):93-102. doi: 10.1097/01.jnr.0000387567.41941.14. PMID 16741859
- [Background] Grocke D. Overview of research in the Bonny Method of Guided Imagery and Music. Voices: A World Forum for Music Therapy, 10(3), 2010
- [Background] Lin MF, Hsu MC, Chang HJ, Hsu YY, Chou MH, Crawford P. Pivotal moments and changes in the Bonny Method of Guided Imagery and Music for patients with depression. J Clin Nurs. 2010 Apr;19(7-8):1139-48. doi: 10.1111/j.1365-2702.2009.03140.x. PMID 20492059
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Maack C, Nolan P. The Effects of Guided Imagery andMusic Therapy on Reported Change in Normal Adults. J Music Ther. 1999;36(1):39-55. doi: 10.1093/jmt/36.1.39. PMID 10519844
- [Background] McKinney CH, Honig TJ. Health Outcomes of a Series of Bonny Method of Guided Imagery and Music Sessions: A Systematic Review. J Music Ther. 2017 Mar 1;54(1):1-34. doi: 10.1093/jmt/thw016. PMID 27941132
- [Background] Rush AJ, Trivedi MH, Carmody TJ, Ibrahim HM, Markowitz JC, Keitner GI, Kornstein SG, Arnow B, Klein DN, Manber R, Dunner DL, Gelenberg AJ, Kocsis JH, Nemeroff CB, Fawcett J, Thase ME, Russell JM, Jody DN, Borian FE, Keller MB. Self-reported depressive symptom measures: sensitivity to detecting change in a randomized, controlled trial of chronically depressed, nonpsychotic outpatients. Neuropsychopharmacology. 2005 Feb;30(2):405-16. doi: 10.1038/sj.npp.1300614. PMID 15578008
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300